CLINICAL TRIAL: NCT04033952
Title: Strategy Training on Improving Executive Functions in Persons Following Acquired Brain Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Feng-Hang Chang, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201905030
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Cognitive Impairment; Stroke; Acquired Brain Injury
Keywords: Stroke; Cognition; Rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Stroke; Brain Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned Interventions (Experimental): The OPASS program will be delivered to the intervention group. The intervention protocols of the OPASS program were developed based on the strategy training guidelines developed by Skidmore et al. and based on the findings identified from the feasibility study. Trained research therapists will take the responsibility for delivering the intervention to participants. The program consists of four critical ingredients: self-selected goals, self-evaluation of performance, strategy development, and implementation, and therapeutic guided discovery.
  Interventions: Behavioral: Strategy Training
- Reflective listening (No Intervention): Participants in the control group will receive dose-matched non-active intervention carried out by a trained research staff. The staff will use scripted questions to provoke participants to describe their experiences and feelings about their disease and their usual-care rehabilitation activities.

INTERVENTIONS:
Behavioral: Strategy Training — This approach is different from traditional direct skill training, which emphasizes clinicians' responsibility on identifying their patients' challenges in performing activities and teaching patients task-specific problem-solving strategies. Strategy training, on the other hand, requires clinicians to take a role as a facilitator, guiding participants to learn through prompts and questions. In the training process, participants learn to develop their own problem-solving strategies and work through the problems they have, through which they can develop self-efficacy and confidence to manage participation challenges. Participants can also generalize the strategies they learn to other similar problems they encounter in daily life.
  Arms: Assigned Interventions

SUMMARY:
About two-third individuals with acquired brain injury (ABI) experience cognitive impairments. Deficits in executive functions is one of the most prevalent cognitive impairments following ABI which result in decline of recovery and independence. Lack of intervention shows evidence of immediate and long-term effect on executive function which is critical after returning to the community. The overall aim of this study is to examine the efficacy of strategy training intervention on executive functions and participation on community-dwelling people with ABI. Findings of the study will provide unequivocal evidence on the duration of effectiveness of strategy training and support the development and application of the program in rehabilitation practice.

DETAILED DESCRIPTION:
The study will use a double-blinded, parallel-group randomized controlled trial to assess the efficacy of the strategy training intervention program in comparison to the control group. The investigators will recruit community-dwelling individuals with ABI in outpatient rehabilitation units and randomly assign them to the intervention group and the control group at a 1:1 ratio. Participants in the intervention group will receive strategy training 2 times per week for 10-15 sessions and participants in the control group will receive dose-matched non-active intervention carried out by a trained therapist. These efforts will allow the investigators to address the gap in rehabilitation research by demonstrating the effectiveness of strategy training on rebuilding and maintaining executive functions and lessening disability. This evidence will be important for rehabilitation practitioners to provide effective treatment to patients with cognitive impairments and will contribute to the improvement of quality of care of rehabilitation services.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20 years and older
* Has a diagnosis of Acquired Brain Injury
* Understand Mandarin
* Has cognitive impairment
* Provide informed consent

Exclusion Criteria:

* Have severe aphasia
* Have a pre-stroke diagnosis of dementia, current major depressive disorder, substance use, or other psychiatric disorders that may impede them from continually participating in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Stroop Test | Change from baseline to post-intervention within 1 week
  Stroop test is a behavioral cognitive assessment tool. Participants will be asked to read out the ink color of the word as accurately and as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time and error to complete the task will be calculated and recorded, in which a longer completion time and more error will indicate poorer outcome. Construct validity of the Stroop Test in the TBI population has been published.
Trail-Making Test (TMT A and B) | Change from baseline to post-intervention within 1 week
  Trail-Making Test (TMT A and B) will be used to measure sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in an ascending order (1-A-2-B-3-C...). The Time and the amount of needed reminders to complete TMT A and B will be calculated, in which a longer completion time and more error will indicate poorer outcome. This instrument was validated in healthy people, patients with head injury, vascular disorders, and other diverse populations.
Montreal Cognitive Assessment (MoCA) | Change from baseline to post-intervention within 1 week
  Montreal Cognitive Assessment (MoCA) is a clinician-reported measure consisting of cognition domains such as: visuospatial skills, executive functions, attention, concentration, calculation, language, abstraction, memory, and orientation. The summary score ranges from 0-30 points with higher scores indicating better cognitive function.

SECONDARY OUTCOMES:
Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms | Change from baseline to post-intervention within 1 week
  The Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms consists of three subscales that assesses three activity domains: basic mobility (18 items), daily activity (15 items), and applied cognitive (19 items). Each item asks the respondent to rate the difficulty to perform specified activities using a 4-point scale. The summary scores range 18-72, 15-60, 19-76 points respectively among three subscales. Higher score indicates better function of the specific domain. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms | Change from post-intervention to 3 month follow-up, within 2 weeks
  The Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms consists of three subscales that assesses three activity domains: basic mobility (18 items), daily activity (15 items), and applied cognitive (19 items). Each item asks the respondent to rate the difficulty to perform specified activities using a 4-point scale. The summary scores range 18-72, 15-60, 19-76 points respectively among three subscales. Higher score indicates better function of the specific domain. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms | Change from 3 month to 6 month follow-up, within 2 weeks
  The Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms consists of three subscales that assesses three activity domains: basic mobility (18 items), daily activity (15 items), and applied cognitive (19 items). Each item asks the respondent to rate the difficulty to perform specified activities using a 4-point scale. The summary scores range 18-72, 15-60, 19-76 points respectively among three subscales. Higher score indicates better function of the specific domain. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms | Change from 6 month to 12 month follow-up, within 2 weeks
  The Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms consists of three subscales that assesses three activity domains: basic mobility (18 items), daily activity (15 items), and applied cognitive (19 items). Each item asks the respondent to rate the difficulty to perform specified activities using a 4-point scale. The summary scores range 18-72, 15-60, 19-76 points respectively among three subscales. Higher score indicates better function of the specific domain. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Healing encounters and attitudes list positive outlook questionnaire short form (HEAL-PO) | Change from baseline to post-intervention within 1 week
  The Healing encounters and attitudes list positive outlook questionnaire short form (HEAL-PO) consists of 6 statements about perceived value on confidence and optimism in general. Each item is ranked on a 1 to 5 Likert-type scale. The summary score ranges from 6-30 points. Higher score indicates a more positive attitude on the participant. Scores are summed and then converted to T-score.
Healing encounters and attitudes list positive outlook questionnaire short form (HEAL-PO) | Change from post-intervention to 3 month follow-up, within 2 weeks
  The Healing encounters and attitudes list positive outlook questionnaire short form (HEAL-PO) consists of 6 statements about perceived value on confidence and optimism in general. Each item is ranked on a 1 to 5 Likert-type scale. The summary score ranges from 6-30 points. Higher score indicates a more positive attitude on the participant. Scores are summed and then converted to T-score.
Healing encounters and attitudes list positive outlook questionnaire short form (HEAL-PO) | Change from 3 month to 6 month follow-up, within 2 weeks
  The Healing encounters and attitudes list positive outlook questionnaire short form (HEAL-PO) consists of 6 statements about perceived value on confidence and optimism in general. Each item is ranked on a 1 to 5 Likert-type scale. The summary score ranges from 6-30 points. Higher score indicates a more positive attitude on the participant. Scores are summed and then converted to T-score.
Healing encounters and attitudes list positive outlook questionnaire short form (HEAL-PO) | Change from 6 month to 12 month follow-up, within 2 weeks
  The Healing encounters and attitudes list positive outlook questionnaire short form (HEAL-PO) consists of 6 statements about perceived value on confidence and optimism in general. Each item is ranked on a 1 to 5 Likert-type scale. The summary score ranges from 6-30 points. Higher score indicates a more positive attitude on the participant. Scores are summed and then converted to T-score.
General Self Efficacy Scale (GSCS) | Change from baseline to post-intervention within 1 week
  The General Self Efficacy Scale is a 10-item scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. Each item is rated using a 1-4 Likert scale, with higher score indicating greater self-efficacy. The summary score ranges from 10-40.
General Self Efficacy Scale (GSCS) | Change from post-intervention to 3 month follow-up, within 2 weeks
  The General Self Efficacy Scale is a 10-item scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. Each item is rated using a 1-4 Likert scale, with higher score indicating greater self-efficacy. The summary score ranges from 10-40.
General Self Efficacy Scale (GSCS) | Change from 3 month to 6 month follow-up, within 2 weeks
  The General Self Efficacy Scale is a 10-item scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. Each item is rated using a 1-4 Likert scale, with higher score indicating greater self-efficacy. The summary score ranges from 10-40.
General Self Efficacy Scale (GSCS) | Change from 6 month to 12 month follow-up, within 2 weeks
  The General Self Efficacy Scale is a 10-item scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. Each item is rated using a 1-4 Likert scale, with higher score indicating greater self-efficacy. The summary score ranges from 10-40.
Canadian Occupational Performance Measure (COPM) | Change from baseline to post-intervention within 1 week
  The Canadian Occupational Performance Measure inquires the client to identify important goals in their daily life and rate their importance, performance and satisfaction for each goal on a 10-point visual analog scale. The summary score ranges from 1-10 on each domain. Higher score indicates a more important, better performance and higher satisfaction on each determined goal. Scores are summed and then converted to T-score for analysis.
Canadian Occupational Performance Measure (COPM) | Change from post-intervention to 3 month follow-up, within 2 weeks
  The Canadian Occupational Performance Measure inquires the client to identify important goals in their daily life and rate their importance, performance and satisfaction for each goal on a 10-point visual analog scale. The summary score ranges from 1-10 on each domain. Higher score indicates a more important, better performance and higher satisfaction on each determined goal. Scores are summed and then converted to T-score for analysis.
Canadian Occupational Performance Measure (COPM) | Change from 3 month to 6 month follow-up, within 2 weeks
  The Canadian Occupational Performance Measure inquires the client to identify important goals in their daily life and rate their importance, performance and satisfaction for each goal on a 10-point visual analog scale. The summary score ranges from 1-10 on each domain. Higher score indicates a more important, better performance and higher satisfaction on each determined goal. Scores are summed and then converted to T-score for analysis.
Canadian Occupational Performance Measure (COPM) | Change from 6 month to 12 month follow-up, within 2 weeks
  The Canadian Occupational Performance Measure inquires the client to identify important goals in their daily life and rate their importance, performance and satisfaction for each goal on a 10-point visual analog scale. The summary score ranges from 1-10 on each domain. Higher score indicates a more important, better performance and higher satisfaction on each determined goal. Scores are summed and then converted to T-score for analysis.
Stroop Test | Change from post-intervention to 3 month follow-up, within 2 weeks
  Stroop test is a behavioral cognitive assessment tool. Participants will be asked to read out the ink color of the word as accurately and as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time and error to complete the task will be calculated and recorded, in which a longer completion time and more error will indicate poorer outcome. Construct validity of the Stroop Test in the TBI population has been published.
Stroop Test | Change from 3 month to 6 month follow-up, within 2 weeks
  Stroop test is a behavioral cognitive assessment tool. Participants will be asked to read out the ink color of the word as accurately and as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time and error to complete the task will be calculated and recorded, in which a longer completion time and more error will indicate poorer outcome. Construct validity of the Stroop Test in the TBI population has been published.
Stroop Test | Change from 6 month to 12 month follow-up, within 2 weeks
  Stroop test is a behavioral cognitive assessment tool. Participants will be asked to read out the ink color of the word as accurately and as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time and error to complete the task will be calculated and recorded, in which a longer completion time and more error will indicate poorer outcome. Construct validity of the Stroop Test in the TBI population has been published.
Trail-Making Test (TMT A and B) | Change from post-intervention to 3 month follow-up, within 2 weeks
  Trail-Making Test (TMT A and B) will be used to measure sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in an ascending order (1-A-2-B-3-C...). The Time and the amount of needed reminders to complete TMT A and B will be calculated, in which a longer completion time and more error will indicate poorer outcome. This instrument was validated in healthy people, patients with head injury, vascular disorders, and other diverse populations.
Trail-Making Test (TMT A and B) | Change from 3 month to 6 month follow-up, within 2 weeks
  Trail-Making Test (TMT A and B) will be used to measure sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in an ascending order (1-A-2-B-3-C...). The Time and the amount of needed reminders to complete TMT A and B will be calculated, in which a longer completion time and more error will indicate poorer outcome. This instrument was validated in healthy people, patients with head injury, vascular disorders, and other diverse populations.
Trail-Making Test (TMT A and B) | Change from 6 month to 12 month follow-up, within 2 weeks
  Trail-Making Test (TMT A and B) will be used to measure sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in an ascending order (1-A-2-B-3-C...). The Time and the amount of needed reminders to complete TMT A and B will be calculated, in which a longer completion time and more error will indicate poorer outcome. This instrument was validated in healthy people, patients with head injury, vascular disorders, and other diverse populations.
National Institutes of Health Stroke scale (NIHSS) | Change from baseline to post-intervention within 1 week
  The National Institutes of Health Stroke scale (NIHSS) is a 15-item measurement designed to assess symptoms indicating severity of stroke by clinicians. Each item is rated 0-2 or 0-3 points according to the symptoms which are commonly seen after stroke . The summary score ranges from 0-42 with higher score indicating greater severity of stroke.
National Institutes of Health Stroke scale (NIHSS) | Change from post-intervention to 3 month follow-up, within 2 weeks
  The National Institutes of Health Stroke scale (NIHSS) is a 15-item measurement designed to assess symptoms indicating severity of stroke by clinicians. Each item is rated 0-2 or 0-3 points according to the symptoms which are commonly seen after stroke . The summary score ranges from 0-42 with higher score indicating greater severity of stroke.
National Institutes of Health Stroke scale (NIHSS) | Change from 3 month to 6 month follow-up, within 2 weeks
  The National Institutes of Health Stroke scale (NIHSS) is a 15-item measurement designed to assess symptoms indicating severity of stroke by clinicians. Each item is rated 0-2 or 0-3 points according to the symptoms which are commonly seen after stroke . The summary score ranges from 0-42 with higher score indicating greater severity of stroke.
National Institutes of Health Stroke scale (NIHSS) | Change from 6 month to 12 month follow-up, within 2 weeks
  The National Institutes of Health Stroke scale (NIHSS) is a 15-item measurement designed to assess symptoms indicating severity of stroke by clinicians. Each item is rated 0-2 or 0-3 points according to the symptoms which are commonly seen after stroke . The summary score ranges from 0-42 with higher score indicating greater severity of stroke.
Rancho Los Amigos Scale-Revised (RLAS-R) | Change from baseline to post-intervention within 1 week
  Rancho Los Amigos Scale-Revised (RLAS-R) is an ordinal scale which describes the cognitive and behavioral patterns found in brain injury patients as they recover from injury. The levels are assessed by clinicians and range from 1 to 10 with higher scores indicating better functioning on brain injury participants.
Rancho Los Amigos Scale-Revised (RLAS-R) | Change from post-intervention to 3 month follow-up, within 2 weeks
  Rancho Los Amigos Scale-Revised (RLAS-R) is an ordinal scale which describes the cognitive and behavioral patterns found in brain injury patients as they recover from injury. The levels are assessed by clinicians and range from 1 to 10 with higher scores indicating better functioning on brain injury participants.
Rancho Los Amigos Scale-Revised (RLAS-R) | Change from 3 month to 6 month follow-up, within 2 weeks
  Rancho Los Amigos Scale-Revised (RLAS-R) is an ordinal scale which describes the cognitive and behavioral patterns found in brain injury patients as they recover from injury. The levels are assessed by clinicians and range from 1 to 10 with higher scores indicating better functioning on brain injury participants.
Rancho Los Amigos Scale-Revised (RLAS-R) | Change from 6 month to 12 month follow-up, within 2 weeks
  Rancho Los Amigos Scale-Revised (RLAS-R) is an ordinal scale which describes the cognitive and behavioral patterns found in brain injury patients as they recover from injury. The levels are assessed by clinicians and range from 1 to 10 with higher scores indicating better functioning on brain injury participants.
Modified Rankin Scale (mRS) | Change from baseline to post-intervention within 1 week
  The modified Rankin Scale (mRS) is designed to measure the degree of disability after a stroke. Each participant is rated 0-6 point on an ordinal scale with higher score indicating greater disability after stroke.
Modified Rankin Scale (mRS) | Change from post-intervention to 3 month follow-up, within 2 weeks
  The modified Rankin Scale (mRS) is designed to measure the degree of disability after a stroke. Each participant is rated 0-6 point on an ordinal scale with higher score indicating greater disability after stroke.
Modified Rankin Scale (mRS) | Change from 3 month to 6 month follow-up, within 2 weeks
  The modified Rankin Scale (mRS) is designed to measure the degree of disability after a stroke. Each participant is rated 0-6 point on an ordinal scale with higher score indicating greater disability after stroke.
Modified Rankin Scale (mRS) | Change from 6 month to 12 month follow-up, within 2 weeks
  The modified Rankin Scale (mRS) is designed to measure the degree of disability after a stroke. Each participant is rated 0-6 point on an ordinal scale with higher score indicating greater disability after stroke.
Euro-QoL-5-Dimension (EQ-5D) | Change from baseline to post-intervention within 1 week
  The Euro-QoL-5-Dimension (EQ-5D) is used to assess participant's health related quality of life which consist of 5 ordinal scale items and 1 item with visual analog scale. Ordinal scales are rated 0-3 points with higher score indicating the pooer health-related quality of life. visual analog scale are rated by respondents reporting perceived health status with a grade ranging from 0 to 100 with higher score indicating the better health status).
Euro-QoL-5-Dimension (EQ-5D) | Change from post-intervention to 3 month follow-up, within 2 weeks
  The Euro-QoL-5-Dimension (EQ-5D) is used to assess participant's health related quality of life which consist of 5 ordinal scale items and 1 item with visual analog scale. Ordinal scales are rated 0-3 points with higher score indicating the pooer health-related quality of life. visual analog scale are rated by respondents reporting perceived health status with a grade ranging from 0 to 100 with higher score indicating the better health status).
Euro-QoL-5-Dimension (EQ-5D) | Change from 3 month to 6 month follow-up, within 2 weeks
  The Euro-QoL-5-Dimension (EQ-5D) is used to assess participant's health related quality of life which consist of 5 ordinal scale items and 1 item with visual analog scale. Ordinal scales are rated 0-3 points with higher score indicating the pooer health-related quality of life. visual analog scale are rated by respondents reporting perceived health status with a grade ranging from 0 to 100 with higher score indicating the better health status).
Euro-QoL-5-Dimension (EQ-5D) | Change from 6 month to 12 month follow-up, within 2 weeks
  The Euro-QoL-5-Dimension (EQ-5D) is used to assess participant's health related quality of life which consist of 5 ordinal scale items and 1 item with visual analog scale. Ordinal scales are rated 0-3 points with higher score indicating the pooer health-related quality of life. visual analog scale are rated by respondents reporting perceived health status with a grade ranging from 0 to 100 with higher score indicating the better health status).
Qualitative data | After intervention, an average of 2 month
  Qualitative in-depth interviews with participants, caregivers, and therapists will be conducted following the intervention. In-depth interviews will be conducted by well-trained interviewers at the end of each participant's intervention. The research team will develop an interview guide consisting of a series of open-ended questions. All intervention sessions will be audio-recorded and transcribed verbatim. Observational data and notes from the therapists, assessors, and research team meetings will be collected and reviewed by the research team throughout the study.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | Change from baseline to post-intervention within 1 week
  The PM-3D4D is a 19-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community. Respondents are asked to rate each item on four dimensions: (1) 'Diversity of participation' (yes [1] vs. no [0]); (2) 'Frequency'(5- and 7-point scales, from "never" to "everyday or almost everyday"); (3) 'Desire for change' (yes [1] vs. no[0]); and (4) 'Perceived difficulty' (4-point scale, from "very difficult" [1] to "not difficult at all" [4]). Each dimensional score of the PM-3D4D can be separately summed for each domain. Psychometric properties of the PM-3D4D were established in rehabilitation populations.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | Change from post-intervention to 3 month follow-up, within 2 weeks
  The PM-3D4D is a 19-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community. Respondents are asked to rate each item on four dimensions: (1) 'Diversity of participation' (yes [1] vs. no [0]); (2) 'Frequency'(5- and 7-point scales, from "never" to "everyday or almost everyday"); (3) 'Desire for change' (yes [1] vs. no[0]); and (4) 'Perceived difficulty' (4-point scale, from "very difficult" [1] to "not difficult at all" [4]). Each dimensional score of the PM-3D4D can be separately summed for each domain. Psychometric properties of the PM-3D4D were established in rehabilitation populations.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | Change from 3 month to 6 month follow-up, within 2 weeks
  The PM-3D4D is a 19-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community. Respondents are asked to rate each item on four dimensions: (1) 'Diversity of participation' (yes [1] vs. no [0]); (2) 'Frequency'(5- and 7-point scales, from "never" to "everyday or almost everyday"); (3) 'Desire for change' (yes [1] vs. no[0]); and (4) 'Perceived difficulty' (4-point scale, from "very difficult" [1] to "not difficult at all" [4]). Each dimensional score of the PM-3D4D can be separately summed for each domain. Psychometric properties of the PM-3D4D were established in rehabilitation populations.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | Change from 6 month to 12 month follow-up, within 2 weeks
  The PM-3D4D is a 19-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community. Respondents are asked to rate each item on four dimensions: (1) 'Diversity of participation' (yes [1] vs. no [0]); (2) 'Frequency'(5- and 7-point scales, from "never" to "everyday or almost everyday"); (3) 'Desire for change' (yes [1] vs. no[0]); and (4) 'Perceived difficulty' (4-point scale, from "very difficult" [1] to "not difficult at all" [4]). Each dimensional score of the PM-3D4D can be separately summed for each domain. Psychometric properties of the PM-3D4D were established in rehabilitation populations.
Resting-state functional Magnetic Resonance Imaging scan (rs-fMRI) | Change from baseline to post-intervention within 1 week
  The Resting-state (rs-fMRI) scan will be administered by a 3T Siemens Magnetom Trio-Tim magnet scanner at National Yang-Ming University. Participants will be asked to keep their eyes closed, heads still, not falling sleep, and think nothing in particular. A T2*-weighted gradient-echo echo planar imaging (EPI) sequence will be employed with TR/TE/FA = 2000 ms/30 ms/90°, 185 time points, resolution: 3×3×3 mm3, 35 axial slides and 6 minutes total scan time. Each participant's relative activity time courses of the blood oxygenation level-dependent (BOLD) response will be collected for analysis.
Resting-state functional Magnetic Resonance Imaging scan (rs-fMRI) | Change from post-intervention to 1 year follow-up, within 2 weeks
  The Resting-state (rs-fMRI) scan will be administered by a 3T Siemens Magnetom Trio-Tim magnet scanner at National Yang-Ming University. Participants will be asked to keep their eyes closed, heads still, not falling sleep, and think nothing in particular. A T2*-weighted gradient-echo echo planar imaging (EPI) sequence will be employed with TR/TE/FA = 2000 ms/30 ms/90°, 185 time points, resolution: 3×3×3 mm3, 35 axial slides and 6 minutes total scan time. Each participant's relative activity time courses of the blood oxygenation level-dependent (BOLD) response will be collected for analysis.
functional Magnetic Resonance Imaging scan with a Color Stroop task | Change from baseline to immediately post-intervention within 1 week
  The functional Magnetic Resonance Imaging scan with a Stroop task will be administered by a 3T Siemens Magnetom Trio-Tim magnet scanner at National Yang-Ming University. A segmented Stroop modified task programmed with E-Prime package will be administered. Participants will be asked to press the corresponding color of the word as accurately and as soon as possible during the task. The ink color of the word could be congruent or incongruent with the written color name. A total scan time is approximately 7 minutes. Specific regions of interest (ROIs), including prefrontal regions will be selected individually for each subject, using a combination of anatomical and functional criteria. The average beta values of the contrast between different levels of task difficulties in these ROIs will be extracted and analyzed.
functional Magnetic Resonance Imaging scan with a Color Stroop task | Change from post-intervention to 1 year follow-up, within 2 weeks
  The functional Magnetic Resonance Imaging scan with a Stroop task will be administered by a 3T Siemens Magnetom Trio-Tim magnet scanner at National Yang-Ming University. A segmented Stroop modified task programmed with E-Prime package will be administered. Participants will be asked to press the corresponding color of the word as accurately and as soon as possible during the task. The ink color of the word could be congruent or incongruent with the written color name. A total scan time is approximately 7 minutes. Specific regions of interest (ROIs), including prefrontal regions will be selected individually for each subject, using a combination of anatomical and functional criteria. The average beta values of the contrast between different levels of task difficulties in these ROIs will be extracted and analyzed.
functional Magnetic Resonance Imaging scan of anatomical structure | Change from baseline to post-intervention within 1 week
  The functional Magnetic Resonance Imaging scan of anatomical structure will be administered by a 3T Siemens Magnetom Trio-Tim magnet scanner at National Yang-Ming University. Participants will be asked to keep their eyes closed, heads still, not falling sleep, and think nothing in particular. A high-resolution three-dimensional MPRAGE sequence will be used to obtain T1-weighted images with 1mm3 isotropic resolution with a scan time of approximately 4.5 min.
functional Magnetic Resonance Imaging scan of anatomical structure | Change from post-intervention to 1 year follow-up, within 2 weeks
  The functional Magnetic Resonance Imaging scan of anatomical structure will be administered by a 3T Siemens Magnetom Trio-Tim magnet scanner at National Yang-Ming University. Participants will be asked to keep their eyes closed, heads still, not falling sleep, and think nothing in particular. A high-resolution three-dimensional MPRAGE sequence will be used to obtain T1-weighted images with 1mm3 isotropic resolution with a scan time of approximately 4.5 min.
functional Magnetic Resonance Imaging scan with a Emotion Stroop task | Change from baseline to post-intervention within 1 week
  The functional Magnetic Resonance Imaging scan with a Stroop task will be administered by a 3T Siemens Magnetom Trio-Tim magnet scanner at National Yang-Ming University. A segmented Stroop modified task programmed with E-Prime package will be administered. Participants will be asked to press the corresponding emotion of the word as accurately and as soon as possible during the task. The word representing the emotion could be congruent or incongruent with the background facial expression. A total scan time is approximately 9.5 minutes. Specific regions of interest (ROIs), including prefrontal regions will be selected individually for each subject, using a combination of anatomical and functional criteria. The average beta values of the contrast between different levels of task difficulties in these ROIs will be extracted and analyzed.
functional Magnetic Resonance Imaging scan with a Emotion Stroop task | Change from post-intervention to 1 year follow-up, within 2 weeks
  The functional Magnetic Resonance Imaging scan with a Stroop task will be administered by a 3T Siemens Magnetom Trio-Tim magnet scanner at National Yang-Ming University. A segmented Stroop modified task programmed with E-Prime package will be administered. Participants will be asked to press the corresponding emotion of the word as accurately and as soon as possible during the task. The word representing the emotion could be congruent or incongruent with the background facial expression. A total scan time is approximately 9.5 minutes. Specific regions of interest (ROIs), including prefrontal regions will be selected individually for each subject, using a combination of anatomical and functional criteria. The average beta values of the contrast between different levels of task difficulties in these ROIs will be extracted and analyzed.
Healing encounters and attitudes list patient-provider connection short form (HEAL-PPC) | At the time of post-intervention within 1 week
  The Patient-Provider Connection Short Form consists of 7 statements in which participants are asked to rate the degree to which they feel the therapist understands and respects them, and provides them with enough information. Each item is ranked on a 1 to 5 Likert-type scale. The total value of the scale ranges from 7 to 35 with a higher score reflecting more positive perspectives a patient had on the connection between patient and health provider. Scores are summed and then converted to T-score.
Montreal Cognitive Assessment (MoCA) | Change from post-intervention to 3 month follow-up, within 2 weeks
  Montreal Cognitive Assessment (MoCA) is a clinician-reported measure consisting of cognition domains such as: visuospatial skills, executive functions, attention, concentration, calculation, language, abstraction, memory, and orientation. The summary score ranges from 0-30 points with higher scores indicating better cognitive function.
Montreal Cognitive Assessment (MoCA) | Change from 3 month to 6 month follow-up, within 2 weeks
  Montreal Cognitive Assessment (MoCA) is a clinician-reported measure consisting of cognition domains such as: visuospatial skills, executive functions, attention, concentration, calculation, language, abstraction, memory, and orientation. The summary score ranges from 0-30 points with higher scores indicating better cognitive function.
Montreal Cognitive Assessment (MoCA) | Change from 6 month to 12 month follow-up, within 2 weeks
  Montreal Cognitive Assessment (MoCA) is a clinician-reported measure consisting of cognition domains such as: visuospatial skills, executive functions, attention, concentration, calculation, language, abstraction, memory, and orientation. The summary score ranges from 0-30 points with higher scores indicating better cognitive function.
Pittsburgh Rehabilitation Participation Scale | During the procedure
  Pittsburgh Rehabilitation Participation Scale is assessed on a 6-point Likert-type scale reflecting the therapists observations of patient participation. The summary score is transformed to an average score for interpretation. The score ranges from 0-6 points with higher scores indicating better participation in each session.
Level of understanding of the intervention session | During the procedure
  Level of understanding of the intervention session is rated by clinicians with a structured questionnaire developed by the research team. A 3 point ordinal scale is administered with a higher score indicating better level of understanding of the intervention session.The total value of the scale depends on the lessons the participant received, ranging from 1*amount of received lessons - 3*amount of received lessons. The score is adopted in the form of average score, ranging from 1 to 3 points.
Healing encounters and attitudes list treatment expectancy short form (HEAL-TE) | baseline, pre-intervention
  Healing encounters and attitudes list treatment expectancy short form is a 6-item self-rated measurement designed to assess the expectations of a participant about whether the treatment will be helpful. Each item will be scored in a 5-point Likert scale. The total value of the scale ranges from 5 to 30 with a higher score indicating higher expectation of the treatment. The score is adopted in the form of average score, ranging from 1 to 5 points.
Client Satisfaction Questionnaire (CSQ) | At the time of post-intervention within 1 week
  Client Satisfaction Questionnaire is a 8 item questionnaire of 4-point Likert scale reflecting the satisfaction of the treatment. The score is adopted in the form of an average score ranging from 1 to 4 points with a higher score indicating higher satisfaction of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Hang Chang, Principal Investigator — Taipei Medical University
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital Bei-Hu branch, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University, Taipei

IPD SHARING:
Plan to Share IPD: No
The IPD is not planned to be shared.